CLINICAL TRIAL: NCT02664779
Title: Determination and Comparison of Short-term Effectiveness of Three Methods Used for Recognition of Arrhythmias in People With Different Degrees of Medical Training (Advanced Life Support Workshop Participants-ALS): Randomized Controlled Educational Experiment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALS1
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arrhythmia diagnosis with the 10 steps method (Experimental): Of participants whom attending the workshop, we will take 84 whom agree to participate and sign the informed consent. They will be divided into subgroups according to their degree of medical training (nursing technicians, university nursing students, university medical students, nurse practitioners graduates, Professional medical graduates, residents of medical specialties and specialists) and randomly assigned one by one from each educational subgroup to 3 intervention groups A, B or C (A = 10 STEPS method, B = 6 STEPS method, C = 4 STEPS method ) so that each group has the third participants of each level of education ensuring matched groups on the level of training of participants in each group. Following this, an equal theoretical test will be performed for all groups to determine the knowledge base in arrhythmias.
  Interventions: Other: Arrhythmia diagnosis with the 10 steps method
- Arrhythmia diagnosis with the 6 steps method (Active Comparator): Of participants whom attending the workshop, we will take 84 whom agree to participate and sign the informed consent. They will be divided into subgroups according to their degree of medical training (nursing technicians, university nursing students, university medical students, nurse practitioners graduates, Professional medical graduates, residents of medical specialties and specialists) and randomly assigned one by one from each educational subgroup to 3 intervention groups A, B or C (A = 10 STEPS method, B = 6 STEPS method, C = 4 STEPS method ) so that each group has the third participants of each level of education ensuring matched groups on the level of training of participants in each group. Following this, an equal theoretical test will be performed for all groups to determine the knowledge base in arrhythmias
  Interventions: Other: Arrhythmia diagnosis with the 6 steps method
- Arrhythmia diagnosis with the 4 steps method (Active Comparator): Of participants whom attending the workshop, we will take 84 whom agree to participate and sign the informed consent. They will be divided into subgroups according to their degree of medical training (nursing technicians, university nursing students, university medical students, nurse practitioners graduates, Professional medical graduates, residents of medical specialties and specialists) and randomly assigned one by one from each educational subgroup to 3 intervention groups A, B or C (A = 10 STEPS method, B = 6 STEPS method, C = 4 STEPS method ) so that each group has the third participants of each level of education ensuring matched groups on the level of training of participants in each group. Following this, an equal theoretical test will be performed for all groups to determine the knowledge base in arrhythmias
  Interventions: Other: Arrhythmia diagnosis with the 4 steps method

INTERVENTIONS:
Other: Arrhythmia diagnosis with the 10 steps method
  Arms: Arrhythmia diagnosis with the 10 steps method
Other: Arrhythmia diagnosis with the 6 steps method
  Arms: Arrhythmia diagnosis with the 6 steps method
Other: Arrhythmia diagnosis with the 4 steps method
  Arms: Arrhythmia diagnosis with the 4 steps method

SUMMARY:
Background: Arrhythmia recognition is a fundamental skill for the provider of advanced life support (ALS). Acquire it is difficult, leading to the birth of systematic methods in an attempt to simplify and optimize, however, it has not compared the effectiveness among the three methods with more evidence among professionals with varying degrees of medical training (ALS Workshop participants).

Objective: To determine and compare the effectiveness of the three most widespread and with more evidence systematic methods (10, 6 and 4 steps) for the recognition of arrhythmias in a short-term and its perceived easiness among ALS workshop participants.

Methods / design: Educational Cuasi experimental trial with pre and post intervention measurement, blind, with randomized allocation, in 84 ALS workshop participants. Three systematic methods to recognize arrhythmias will be taught and their effectiveness to diagnose in a short-term and its perceived easiness will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* • Health professionals

  * Attend a course in Advanced Life Support in Cali (Colombia), during the study period.
  * Voluntarily accept to participate in the study

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
percentage of subjects who achieve scores greater than or equal to 30 | 15 minutes after delivered the intervention
  For comparison of the percentage of subjects who achieve scores greater than or equal to 30 (approving minimum score) in the practical test of arrhythmia's diagnosis, the test will be the Chi-square (X2), which allows to compare proportions in more than two groups; or Fisher's exact test, submitted that one of the expected values is less than 5.

SECONDARY OUTCOMES:
change in the average scores in the groups | 15 minutes after delivered the intervention
  In order to compare the magnitude of the change in the average scores in the groups trained with each of the 3 methods, both in the the theoretical and practical test of diagnosis of arrhythmias; ANOVA or Mann-Whitney's U, according to the distribution of variables was performed. These comparisons are made to the post intervention measurements and Bonferroni correction for alpha according to the number of comparisons will perform. The analysis of the collected data will be using STATA 10.0 software.

CONTACTS AND LOCATIONS:
Locations (1):
- Cruz Roja Colombiana, Cali, Valle del Cauca Department, Colombia